CLINICAL TRIAL: NCT07137741
Title: The Effect of Family-Integrated Care Based on Swanson's Theory of Caring on Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yongkang Maternal and Child Health Hospital (Other)
Responsible Party: Principal Investigator, huijie zhu, chief nurse, Yongkang Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YongkangMCHH
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Premature Infants
Keywords: Family Integrated Care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): traditional model of hospital care
- FICare nursing method guided by Swanson's caring theory (Experimental): encompasses the following five dimensions: Understanding: A neonatologist provided a comprehensive explanation regarding the developmental progress of premature infants, potential complications, and essential aspects of nursing care to ensure the family gained a thorough understanding of the care requirements for premature infants.
  Accompaniment: Two nursing guides provided essential support to parents of newborns in the NICU, helping to alleviate the anxiety and sense of helplessness among family members and fostering a relationship of trust between the medical staff and the families.
  Help: A neonatal nurse played a guiding role in facilitating parental involvement in the daily care of premature infants, which encompassed feeding guidance, introduction of complementary foods, skin care, and related aspects.
  Empowerment: A psychological counselor was assigned to provide psychological counseling and guidance to new parents, offering appropriate emotional support and assisting them in a
  Interventions: Behavioral: FICare nursing method guided by Swanson's caring theory

INTERVENTIONS:
Behavioral: FICare nursing method guided by Swanson's caring theory — encompasses the following five dimensions: Understanding: A neonatologist provided a comprehensive explanation regarding the developmental progress of premature infants, potential complications, and essential aspects of nursing care to ensure the family gained a thorough understanding of the care requirements for premature infants.
  Accompaniment: Two nursing guides provided essential support to parents of newborns in the NICU, helping to alleviate the anxiety and sense of helplessness among family members and fostering a relationship of trust between the medical staff and the families.
  Help: A neonatal nurse played a guiding role in facilitating parental involvement in the daily care of premature infants, which encompassed feeding guidance, introduction of complementary foods, skin care, and related aspects.
  Empowerment: A psychological counselor was assigned to provide psychological counseling and guidance to new parents, offering appropriate emotional support and assisting them in ac
  Arms: FICare nursing method guided by Swanson's caring theory

SUMMARY:
Previous studies have demonstrated that the implementation of FICare in single-family neonatal units is associated with a reduced risk of late-onset sepsis among preterm infants, a shorter hospital length of stay, a lower risk of rehospitalization, and improved breastfeeding rates.However, the impact of FICare, guided by Swanson's caring theory, on the growth and development of newborns, as well as on parental anxiety and their sense of parenting competence, remains unclear. To address this gap, the investigators conducted a cohort study to investigate these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ranging from 28 to 36 weeks
* stable vital signs for at least 24 hours
* parental accompaniment of preterm infants during hospitalization

Exclusion Criteria:

* preterm infants with severe congenital or genetic disorders
* preterm infants with dysfunction of vital organs
* preterm infants requiring mechanical life support
* preterm infants requiring surgical intervention
* preterm infants with a birth weight below 500 grams

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
head circumference | 6 months
  To measure a preterm infant's head circumference: use a soft tape, wrap snugly over supraorbital ridges and occipital protuberance, read to 0.1cm, repeat twice, record.
body weight | 6 months
  To measure a preterm infant's weight: place on a calibrated, zeroed electronic scale (nappy only), ensure stillness, read to 0.1g, repeat twice, record with date/time.
body length | 6 months
  To measure a preterm infant's length: extend body, align head/heel, use a length board, read to 0.1cm, repeat, record.
STAI scores | 6 months
  STAI (State-Trait Anxiety Inventory) scores assess anxiety levels via two scales: State Anxiety (S-AI) measures temporary anxiety, Trait Anxiety (T-AI) assesses general anxiety proneness.
  Each has 20 items, rated 1-4. Scores range 20-80; higher scores indicate greater anxiety. S-AI ≥40 suggests significant state anxiety; T-AI ≥40 may indicate trait anxiety.
PSOC scores | 6 months
  PSOC (Parenting Sense of Competence Scale) scores assess parental self-efficacy and satisfaction. It has 17 items, rated 1-6, covering efficacy (confidence) and satisfaction (emotional engagement). Scores range 17-102; higher scores mean stronger. parenting competence.

CONTACTS AND LOCATIONS:
Locations (1):
- Yongkang maternal and Child Health Hospital, Guli, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT07137741/Prot_SAP_002.pdf
  • Informed Consent Form (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT07137741/ICF_001.pdf